CLINICAL TRIAL: NCT03637738
Title: Medico Economic Study, Randomized, Comparing Intraoperative Radiotherapy With Intrabeam® on Surgical Resection Bed Versus Conventional Surgery + EBRT in Postmenopausal Patients Operated by Conservative Surgery for Low Risk Breast Cancer
Brief Title: Medico Economic Study, Comparing Intrabeam® on Surgical Resection Bed to Conventional Surgery + EBRT, in Breast Cancer
Acronym: RIOP-SEIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICO-2012-03
Record Dates: First submitted 2018-08-14; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Menopausal Patients; Low-risk Breast Cancer
Keywords: Intrabeam®; intraoperative radiation therapy; conventional external radiotherapy; conservative surgery

STUDY DESIGN:
Intervention Model Description: Medico-economic, National Multicentric, Prospective, Randomized, Comparative, Open study of a medical device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIOP-Intrabeam® system (Experimental): Surgery with Intrabeam®. A first visit will be scheduled at 2 months from surgery then at 6 months then every 6 months for 5 years, then every year after 5 years.
  Additional EBRT may be performed +/- chemotherapy if the treatment received is insufficient.
  Interventions: Radiation: RIOP-Intrabeam® system
- conventional surgery +RTE (Active Comparator): surgery, EBRT over 33 sessions then visit at 6 months then every 6 months 6 for 5 years, then every year after 5 years.
  Interventions: Radiation: conventional surgery +RTE

INTERVENTIONS:
Radiation: RIOP-Intrabeam® system — The radiation source is inserted at the immediately on surgical resection bed after tumorectomy and started for 20 to 55 minutes to perform intraoperative radiotherapy precisely targeting the tissues that present the greatest risk of local recurrence. The applied dose will be 20 Gy on the applicator surface.
  Arms: RIOP-Intrabeam® system
Radiation: conventional surgery +RTE — Conventional EBRT, 5 to 10 weeks after surgery, according to the usual recommendations, 2 Gy per session, 5 sessions per week, with a total dose on the mammary gland of 50 Gy + a boost of 16 Gy on surgical resection bed .
  Arms: conventional surgery +RTE

SUMMARY:
Current breast cancer treatment is based on surgery, radiation, chemotherapy and hormonotherapy. Conservative surgery or mastectomy are followed by complementary externe radiotherapy.

This adjuvant external breast radiotherapy (EBRT) is heavy, spread over more than 6 weeks with :

* 25 sessions and delivery of a unit dose of 2 Gy to obtain a total dose of 50 Gy (5 sessions per week in general);
* 16 Gy overimpression (boost) dose located in the tumour bed, in 5 to 8 fractions, in situations at high risk of recurrence.

In addition, EBRT is responsible for many adverse effects, some of which can lead to lasting or permanent sequelae.

Many focused partial breast irradiation techniques have been developed in recent years with the objective of reducing the duration and morbidity of overall breast irradiation.

Among these techniques, intraoperative breast radiotherapy (IBRT) is recommended in cancers diagnosed at early stages for which tumorectomy is expected and which present a low risk of recurrence.

The main advantages of IBRTare :

* Improvement of the quality of life due to a single session of radiotherapy associated with surgical ;
* Increased precision to deliver the necessary dose in tumour tissue;
* Preservation of surrounding healthy tissue ;
* Reduction in the overall cost of treatment through shorter hospital stays and the absence of medical transport for conventional radiotherapy sessions.

RIOP SEIN is a project supported by Institut National du Cancer (INCa)

, which consists of a medico-economic evaluation of IBRT, with Intrabeam® system on surgical resection bed relative to conventional surgery + EBRT in postmenopausal patients operated by conservative surgery for Low risk breast cancer

DETAILED DESCRIPTION:
Main objective is the economic comparison Intrabeam® system versus EBRT, in terms of real costs. Costs will be taken into account:

* of equipment,
* of staff,
* of transport.

Secondary objectives are :

* Compare local-regional survival without recurrence with conventional irradiation
* Analyze the rate of early and late complications
* Impact of intraoperative irradiation on the esthetic outcome and quality of life of patients

Schedule of the visits :

RIOP arm : Surgery with Intrabeam®. A first visit will be scheduled at 2 months from surgery then at 6 months then every 6 months for 5 years, then every year after 5 years.

RTE arm: surgery, EBRT over 33 sessions then visit at 6 months then every 6 months 6 for 5 years, then every year after 5 years.

In RIOP ARM, additional EBRT may be performed +/- chemotherapy if the treatment received is insufficient.

Quality of life will be assessed in each treatment arm at inclusion before randomization, 2 months after surgery, every 6 months for 5 years and every year after 5 years using quality of life questionnaires: Euroqol EQ 5D, European Organisation for Research and Treatment of Cancer (EORTC)-QlQ-C30 and BR23 module specific for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven invasive ductal breast cancer,
* Menopausal women at least 55 years old,
* Clinical and ultrasound size ≤ to 20 mm, N0,
* Biopsy with all following criteria: SBR I or II, HER2 (0, +, ++ with FISH or SISH required), positive estrogen receptors, no embolus
* No personal history of breast cancer or BRCA gene mutation.
* Social insurance
* Signed consent

Exclusion Criteria:

* Bifocal or bilateral breast cancer,
* Presence of invasive ductal carcinoma with diffuse micro calcifications on mammography,
* Invasive lobular carcinoma,
* Presence of lymph node involvement,
* History of malignant disease if life expectancy without recurrence at 10 years <90%,
* Adult under guardianship,
* History of chest radiation therapy (Hodgkin's).

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2012-06; Primary Completion 2014-08 (Actual); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Actual cost | 2 months after the end of radiotherapy
  Actual cost measured individually for each patient for both techniques used, involving all costs from surgery to 2 months after the end of radiotherapy including costs related to possible acute complications of radiotherapy

SECONDARY OUTCOMES:
Local-regional recurrence rate | 10 years
  Analysis of the local-regional relapse rate with Intrabeam system as compared with the results published with EBRT
Complication rates | 10 years
  Early and late complication rates
Esthetic result | 10 years
  Taking photos at inclusion, 2 months, 1 year, 5 years and 10 years from the end of radiotherapy
quality of life after surgery and radiotherapy | 10 years
  questionnaires EQ 5D
quality of life after surgery and radiotherapy | 10 years
  questionnaires EORTC-QLQ-C30
quality of life after surgery and radiotherapy | 10 years
  questionnaires BR23

CONTACTS AND LOCATIONS:
Overall Officials: MAGALI LE BLANC, MD, Principal Investigator — ICO NANTES
Locations (8):
- France (8):
  - Institut Bergonié, Bordeaux
  - Chu Morvan, Brest
  - Centre G F Leclerc, Dijon
  - Centre Léon Berard, Lyon
  - Institut Paoli Calmette, Marseille
  - INSTITUT REGIONAL DU CANCER MONTPELLIER - Val D'Aurelle, Montpellier
  - Hôpital Saint Louis, Paris
  - Centre René Gauducheau, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No